CLINICAL TRIAL: NCT02113397
Title: Comparative Evaluation of Bacterial Diversity and Richness in CF Lung in Patients Who Use Cycled Every Other Month Tobramycin Inhalation Powder (TOBI™ Podhaler™) Or Continuous Alternating Therapy With Tobramycin Inhalation Powder (TOBI™ Podhaler™) and Inhaled Colistimethate
Brief Title: Evaluation of Inhaled Antibiotics on Bacterial Diversity and Richness in the Cystic Fibrosis Lung
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Alex H. Gifford, Assistant Professor of Medicine, Dartmouth-Hitchcock Medical Center
Other Study IDs: D14010; CTBM100DUS02T (Other Grant/Funding Number: Novartis Pharmaceuticals)
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Microbiome; Sputum; Tobramycin; Colistimethate
MeSH Terms: conditions — Cystic Fibrosis | interventions — colistinmethanesulfonic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial genomic DNA will be extracted and purified from sputum samples and sequenced by 454 pyrosequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Continuous Therapy: TOBI™ Podhaler™ 112 mg inhaled by mouth twice daily for 30 days followed by a 30-day cycle colistimethate 75 mg inhaled two times daily. Repeat cycle.
  Interventions: Drug: TOBI™ Podhaler™ 112 mg inhaled twice daily; Drug: Colistimethate 75 mg inhaled two times daily
- Cyclic therapy: TOBI™ Podhaler™ 112 mg inhaled by mouth twice daily for 30 days followed by a 30-day period during which no inhaled antibiotics are used. Repeat cycle.
  Interventions: Drug: TOBI™ Podhaler™ 112 mg inhaled twice daily

INTERVENTIONS:
Drug: TOBI™ Podhaler™ 112 mg inhaled twice daily
  Other Names: Tobramycin inhalation powder
Drug: Colistimethate 75 mg inhaled two times daily
  Groups: Continuous Therapy

SUMMARY:
The purpose of this study is to characterize bacterial diversity and richness in the sputum of cystic fibrosis patients treated with every-other-month TOBI™ Podhaler™ and continuous alternating therapy with TOBI™ Podhaler and colistimethate (Colistin).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis confirmed by mutation analysis of the cystic fibrosis transmembrane conductance regulator gene
* Sputum or throat swab culture positive for Pseudomonas aeruginosa at or within 6 months of enrollment
* Age ≥12 years
* Forced expiratory volume in one second (FEV1) 25-90 percent-predicted

Exclusion Criteria:

* Age <18 years
* Inability to routinely expectorate sputum without induction by hypertonic saline
* Inability to provide or withdrawal of written informed consent
* History of aminoglycoside sensitivity or adverse reaction to inhaled antibiotics
* Serum creatinine ≥ 2.0 mg/dl
* Serum blood urea nitrogen (BUN) ≥40 mg/dl
* Pregnancy or lactating at screening
* History of systemic intravenous anti-Pseudomonal antibiotics within 28 days of enrollment

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with cystic fibrosis who are followed at Dartmouth-Hitchcock Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Simpson Diversity Index | 6 months
  The primary estimate in our study is the mean effects of Continuous Alternating Therapy compared to Cyclic therapy on Simpson Diversity Index (SDI) averaged at month 6

SECONDARY OUTCOMES:
Bacterial Relative Abundance | 6 months
  Using 454 pyrosequencing and quantitative polymerase chain reaction (qPCR) techniques, the relative abundance of various bacterial genera will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Filkins LM, Hampton TH, Gifford AH, Gross MJ, Hogan DA, Sogin ML, Morrison HG, Paster BJ, O'Toole GA. Prevalence of streptococci and increased polymicrobial diversity associated with cystic fibrosis patient stability. J Bacteriol. 2012 Sep;194(17):4709-17. doi: 10.1128/JB.00566-12. Epub 2012 Jun 29. PMID 22753064
- [Background] Price KE, Hampton TH, Gifford AH, Dolben EL, Hogan DA, Morrison HG, Sogin ML, O'Toole GA. Unique microbial communities persist in individual cystic fibrosis patients throughout a clinical exacerbation. Microbiome. 2013 Nov 1;1(1):27. doi: 10.1186/2049-2618-1-27. PMID 24451123